CLINICAL TRIAL: NCT01824030
Title: FFR or OCT Guidance to RevasculariZe Intermediate Coronary Stenosis Using Angioplasty
Acronym: FORZA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Francesco Burzotta, MD, PhD, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6261/13
Record Dates: First submitted 2013-03-28; First posted 2013-04-04 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Ischemic Heart Disease
Keywords: FFR, OCT, Seattle Angina Questionnaire
MeSH Terms: conditions — Myocardial Ischemia; Ornithine Carbamoyltransferase Deficiency Disease

ARMS (2):
- FFR guided PCI arm (Active Comparator): Patients with angiographic intermediate coronary artery stenosis randomized to FFR assessment. PCI performed only if FFR ≤ 0.80
  Interventions: Device: FFR guided PCI
- OCT guided PCI arm (Active Comparator): Patients with angiographic intermediate coronary artery stenosis randomized to OCT. PCI will be performed if:
  1. percentage area stenosis ≥75 %
  2. percentage area stenosis between 50 and 75% and minimal lumen area <2.5 mm2
  3. percentage area stenosis between 50 and 75% and major plaque ulceration
  Interventions: Device: OCT guided PCI

INTERVENTIONS:
Device: FFR guided PCI — FFR to assess coronary artery stenosis severity and indication to perform and eventually optimize percutaneous coronary intervention
  Arms: FFR guided PCI arm
Device: OCT guided PCI — OCT to assess coronary artery stenosis severity and indication to perform and eventually optimize percutaneous coronary intervention
  Arms: OCT guided PCI arm

SUMMARY:
Whether to revascularize patients with angiographically-intermediate coronary lesions (AICL) is a major clinical issue. Intravascular techniques (assessing either the anatomy or the functional effect of coronary stenoses) are routinely used to better characterize coronary lesions. Among these,fractional flow reserve (FFR) provides validated functional insights while optical coherence tomography (OCT) provides high resolution anatomic imaging. Both techniques may be applied to guide decisions regarding the opportunity to revascularize patients with AICL and to optimize the result of percutaneous coronary intervention (PCI). We aim to compare the clinical and the economical impact of FFR versus OCT guidance in the percutaneous management of patients with AICL.

ELIGIBILITY:
Inclusion Criteria:

* single vessel disease with an intermediate coronary artery stenosis
* multivessel disease with multiple intermediate coronary artery stenosis only
* multivessel disease with already treated angiographically critical stenosis and at least one intermediate coronary artery stenosis

Exclusion Criteria:

* age <18 years or impossibility to give informed consent,
* female sex with child-bearing potential,
* life expectancy of less than 12 months or factors making clinical follow-up difficult (no fixed address, etc),
* poor cardiac function as defined by left ventricular global ejection fraction ≤ 30%
* recent (< 7 days) ST-segment elevation myocardial infarction
* recent (< 48 hours) Non ST-segment elevation myocardial infarction
* prior ST-segment elevation myocardial infarction in the territory supplied by the vessel with the intermediate stenosis under investigation
* severe myocardial hypertrophy (interventricular septum thickness > 15 mm, ECG Sokolow's criteria fulfilled)
* severe valvular heart disease
* significant platelet count alteration (<100,000 cells/mm3 or > 700,000 cells/mm3)
* gastrointestinal bleeding requiring surgery or blood transfusions within 4 previous weeks
* history of clotting pathology
* known hypersensitivity to aspirin, heparin, contrast dye
* advance renal failure with glomerular filtration rate < 30 ml/min
* lesions in coronary artery bypass grafts
* multivessel disease requiring coronary aortic bypass graft intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of angina defined as Seattle Angina Questionnaire score < 90 in angina frequency scale, at 13 month follow up from index procedure* | 13 months
  *In case of MACE rate absolute difference of >1% between the two study arms, the primary end-point will be: "Occurrence of Major Cardiovascular Event and angina defined as Seattle Angina Questionnaire score < 90 in angina frequency scale, at 13 months follow up from index procedure"

SECONDARY OUTCOMES:
Occurrence of Major Cardiovascular Event and angina defined as Seattle Angina Questionnaire score < 90 in angina frequency scale, at 13 months follow up from index procedure | 13 months

OTHER OUTCOMES:
Periprocedural costs | 30 days
Periprocedural costs | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Burzotta, MD, PhD, Principal Investigator — Università Cattolica del Sacro Cuore, Roma
Locations (1):
- Policlinico A. Gemelli. Università Cattolica del Sacro Cuore, Rome, Italy

REFERENCES:
- [Derived] Aurigemma C, Ding D, Tu S, Li C, Yu W, Li Y, Leone AM, Romagnoli E, Vergallo R, Maino A, Trani C, Wijns W, Burzotta F. Three-Year Clinical Impact of Murray Law-Based Quantitative Flow Ratio and OCT- or FFR-Guidance in Angiographically Intermediate Coronary Lesions. Circ Cardiovasc Interv. 2024 May;17(5):e013191. doi: 10.1161/CIRCINTERVENTIONS.123.013191. Epub 2024 Apr 25. PMID 38660794
- [Derived] Ding D, Tu S, Li Y, Li C, Yu W, Liu X, Leone AM, Aurigemma C, Romagnoli E, Vergallo R, Trani C, Wijns W, Burzotta F. Quantitative flow ratio modulated by intracoronary optical coherence tomography for predicting physiological efficacy of percutaneous coronary intervention. Catheter Cardiovasc Interv. 2023 Jul;102(1):36-45. doi: 10.1002/ccd.30681. Epub 2023 May 12. PMID 37172214
- [Derived] Burzotta F, Leone AM, Aurigemma C, Zambrano A, Zimbardo G, Arioti M, Vergallo R, De Maria GL, Cerracchio E, Romagnoli E, Trani C, Crea F. Fractional Flow Reserve or Optical Coherence Tomography to Guide Management of Angiographically Intermediate Coronary Stenosis: A Single-Center Trial. JACC Cardiovasc Interv. 2020 Jan 13;13(1):49-58. doi: 10.1016/j.jcin.2019.09.034. PMID 31918942
- [Derived] Leone AM, Burzotta F, Aurigemma C, De Maria GL, Zambrano A, Zimbardo G, Arioti M, Cerracchio E, Vergallo R, Trani C, Crea F. Prospective Randomized Comparison of Fractional Flow Reserve Versus Optical Coherence Tomography to Guide Revascularization of Intermediate Coronary Stenoses: One-Month Results. J Am Heart Assoc. 2019 Aug 6;8(15):e012772. doi: 10.1161/JAHA.119.012772. Epub 2019 Jul 23. PMID 31331219
- [Derived] Burzotta F, Leone AM, De Maria GL, Niccoli G, Coluccia V, Pirozzolo G, Saffioti S, Aurigemma C, Trani C, Crea F. Fractional flow reserve or optical coherence tomography guidance to revascularize intermediate coronary stenosis using angioplasty (FORZA) trial: study protocol for a randomized controlled trial. Trials. 2014 Apr 23;15:140. doi: 10.1186/1745-6215-15-140. PMID 24758510